CLINICAL TRIAL: NCT05280834
Title: Investigation of the Relationship Between Sociodemographic Characteristics and Sexual Health Behaviours of University Students
Brief Title: Investigation of the Sociodemographic Characteristics and Sexual Health Behaviours of University Students
Status: Completed | Type: Observational
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Esra Demirarslan, Instructor Dr., Kastamonu University
Other Study IDs: 80404136-044-E-50015
Record Dates: First submitted 2021-12-02; First posted 2022-03-15 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Sexually Transmitted Diseases
Keywords: students; sexual activities; sexually transmitted diseases; sexual health; community health education
MeSH Terms: conditions — Sexually Transmitted Diseases; Sexual Behavior; Health Education

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The 10-19 age group is defined as the "Adolescent" and the 15-24 age group is defined as the "Youth" by the WHO. Adolescent period is the most vulnerable time to risks in terms of sexual health. Among the sexual health problems experienced by adolescents are sexually transmitted infections(STI), unwanted pregnancies, induced abortions and related complications, not using contraception, STI-induced cancer and infertility, sexual dysfunction.University students are at risk for sexual health because they are in the adolescent age group, they are inexperienced in gaining life experiences, and they are mostly away from the family environment for the first time. Insufficient knowledge in terms of sexual health and insufficient education on sexuality can affect students' attitudes and behaviors related to sexuality. In addition, in developing countries such as Turkey, sexuality is seen as a taboo, and the meanings attributed to sexuality vary according to men and women. In limited studies, it was determined that 24.1% of university student had sexual intercourse at least once, and 40.7% of them had sexual intercourse with more than one person in the last six months. It was determined that 15.5% of the adolescents 60.7% of the youth had sexual experience. In another study with men, it was determined that the students had their first sexual experience at the age of 17-18 on average and 31.0% of them still had active sexual lives. According to the results of a research conducted on first year students of eight universities; It was determined that 19% of the students had sexual experience. These results reveal that one out of every three young people in our country has sexual experience, and that the majority of them are not protected and there is a lack of information about sexuality. It is noteworthy that the rate of becoming sexually active in adolescents and young people is increasing. For this reason, studies are needed to examine the relationship between the status of having a sexual partner and sexual health in university students who have sexual experience. It is important to investigate this relationship and to provide at-risk students with trainings that increase their awareness of sexual health and sexual education. It is planned to examine the relationship between the status of having a sexual partner and sexual health of students studying at Kastamonu University.

DETAILED DESCRIPTION:
Adolescence is the period of life between childhood and adulthood, between the ages of 10 and 19. This period is a unique stage of human development in which the foundations of physical, sexual, and psychosocial development are laid. Adolescents make up one sixth of the world's population. Approximately 85-90% of adolescents, who make up 18% of the entire world population, live in developing countries, including Turkey. The transition from adolescence to adulthood is a complex and exciting period for young adults as they begin to explore their sexual identity and sexual relationships. When starting college, students gain more autonomy over their behaviour and responsibilities related to their health. As a result of this newly acquired autonomy, students frequently engage in various risky behaviours and endanger their health.

Early sexual activity, which is one of the risky health behaviours among adolescents, is increasing worldwide. Various studies conducted in sub-Saharan Africa show that the initiation of premarital sexual intercourse is high among adolescents and this rate is increasing gradually. In a study conducted in North Carolina, it was determined that the first sexual intercourse age of adolescents was 16.5 and 66% of adolescents who had sexual intercourse were between the ages of 15-20. Mohammadi et al. (2006) reported that in their study in Iran 28% of youth aged 15-18 years had at least one sexual intercourse (including hugging, kissing, and any sexual experience from touching to sexual intercourse. In our country, it has been determined that 36.7% of university students have sexual experience and sexual experience is more common in men .

University students are among the population with the highest risk of sexually transmitted infections, unwanted pregnancy and other adverse health outcomes. Young people who are sexually active are exposed to risks such as sexually transmitted diseases and unwanted pregnancies, as their developmental status is insufficient in the assessment and management of these risks. Evidence suggests that young adults aged 20 to 24 are more susceptible to STIs than other age groups. In addition, adolescents are vulnerable to sexually transmitted diseases and infections, including HIV/AIDS, unplanned premature birth, and unsafe abortions as a result of early sexual intercourse due to their limited knowledge of their bodies and sexuality. Halcón, et al. (2001) found benign cellular changes in 15.6%, reactive changes in 9.2%, and epithelial cell abnormalities in 9.9% of adolescent girls who started sexual intercourse at an early age.

The age of first sexual experience decreases in adolescents, contraceptive use also decreases. As the result of non contraception, pregnancy rates were 22.3 per 1,000 women aged 15-19 years and 43% for women aged 18-19 years between 2007 and 2015, birth rates fell 54% for females aged 15-17 years. More than one third of all adolescent girls do not use any contraceptive method during the first sexual intercourse. In a study conducted in Tanzania, it was reported that 29.7% of adolescent boys and 40.3% of adolescent girls did not use contraceptive methods during sexual intercourse. Not using contraceptive methods may cause adolescent pregnancies.

In adolescent pregnancies, the risk of experiencing problems such as preterm labour, perinatal death, fetal and neonatal death, and low birth weight baby is high. However, depression symptoms and deterioration in self-image are more common in young people who start sexual intercourse at a young age. It is noteworthy that the rate of becoming sexually active in adolescents and young people, who make up approximately 20% of the population of our country, is increasing. For this reason, studies are needed to examine the relationship between having a sexual partner and sexual health in university students who have sexual experience. It is thought that it will be important to investigate this relationship and to provide at-risk students with trainings that increase their awareness of sexual health and sexual education. With the results obtained, it is aimed to provide individuals with the necessary motivation, knowledge, and behavioural skills to determine the sexual health problems of the students and to prevent their problems and to improve their sexual health.

Materials and methods:

Participants This cross-sectional study was conducted at 5 faculties and three vocational schools of a university. The population of the research consisted of 13420 undergraduate students studying at faculties and vocational schools. Students who attended the university during the study period and were willing to participate in the study were included in the sample. The minimum sample size of the study was determined according to the frequency formula in cases with a known population. The frequency of the investigated event was accepted as 37% according to the related literature. In conclusion, this study aimed to include 307 students with a minimum sample size for 0.05 deviation and 95% confidence interval (α = 0.05). A total of 825 students participated in the research.

Setting The research was carried out in a university located in the Western Black Sea region, within two weeks (4 weeks in total) when the final exams were held in the 2019 spring and 2020 fall semesters.

Data collection tools In the data collection, a semi-structured interview form was used to determine the sociodemographic characteristics and sexual health behaviours prepared by the researchers in line with the literature.

Data Collection The questionnaire and semi-structured interview form were applied to the students during the 2019-2020 academic year fall semester and spring semester final exams. Question papers were distributed to the students by the researchers in a sealed envelope before the exam time. After the students who volunteered to participate in the research filled out the forms, they submitted them to the researchers in a closed envelope. The practice started on the first day of the exams and continued until the last day.

Ethical dimension of research Before starting the research, permission was obtained from the Non-Interventional Clinical Research Ethics Committee of Karabük University (decision no. 12/1 dated 03.12.2018) and the rectorate of the university where the research would be conducted (approval of the rectorate dated 12.12.2018 and numbered 80404136-044-E-50015). Written informed consent was obtained from the students who volunteered to participate in the study. Throughout the study, the Helsinki Declaration was acted upon. Participants/non-participants did not have any gains/losses such as money, grades, absentee rights, etc.

Statistical analysis:

While evaluating the data, descriptive statistical methods (Number, Percentage, Mean, Standard deviation, variance) were used. The conformity of the data to the normal distribution was determined by the Kruskall-Wallis test in independent samples. and Kendall's Tau-C correlation coefficient was calculated for correlation analyzis.

ELIGIBILITY:
Inclusion Criteria:

* Who wants to be in

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students of a university
Sampling Method: Probability Sample
Enrollment: 825 (Actual)
Dates: Start 2019-12-28 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
age at first sexual intercourse | through study completion, an average of 1 year
  age at first intercourse ill be defined.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander KA, Jemmott LS, Teitelman AM, D'Antonio P. Addressing sexual health behaviour during emerging adulthood: a critical review of the literature. J Clin Nurs. 2015 Jan;24(1-2):4-18. doi: 10.1111/jocn.12640. Epub 2014 Jul 3. PMID 24988875
- [Background] (CDC), C. f. D. C. a. P. (2017). STDs in Adolescents and Young Adults - 2016 STD Surveillance Report. . Retrieved from https://www.cdc.gov/std/life-stages-populations/adolescents-youngadults.htm